CLINICAL TRIAL: NCT01906671
Title: Plasma Kinetics of Tablet and Liquid Formulations of 6-mercaptopurine in Childhood Acute Lymphoblastic Leukemia.
Brief Title: Study on Two Different Formulations of 6-mercaptopurine. Tablet Versus Oral Liquid
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kjeld Schmiegelow (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Sponsor-Investigator, Kjeld Schmiegelow, Professor in Pediatrics and Pediatric Oncology, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 6-MP formulation; 2013-001236-21 (EudraCT Number)
Record Dates: First submitted 2013-07-16; First posted 2013-07-24 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Acute Lymphoblastic Leukemia; 6-mercaptopurine Therapy
Keywords: 6-mercaptopurine; Drug formulation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Puri-Nethol (Experimental): Tablet formulation of 6-mercaptopurine
  Interventions: Drug: Xaluprine; Drug: Puri-Nethol
- Xaluprine (Experimental): Oral liquid formulation of 6-mercaptopurine
  Interventions: Drug: Xaluprine; Drug: Puri-Nethol

INTERVENTIONS:
Drug: Xaluprine — Comparison of plasma kinetics after administration of 6-mercaptopurine in the form of a tablet (Puri-Nethol) and in the form of an oral liquid formulation (Xaluprine). Each patient will be included in both arms of the study, because of the cross-over design.
Drug: Puri-Nethol — Comparison of plasma kinetics after administration of 6-mercaptopurine in the form of a tablet (Puri-Nethol) and in the form of an oral liquid formulation (Xaluprine). Each patient will be included in both arms of the study, because of the cross-over design.

SUMMARY:
Acute lymphoblastic leukemia (ALL) accounts for 30 % of all childhood malignancies. The patients undergo four phases of treatment, finishing with a late maintenance phase in which 6-mercaptopurine and Methotrexate are essential components. Insufficient treatment intensity in this phase is associated with increased risk of relapse. Excessive variation in the bioavailability of 6-mercaptopurine has been observed which can cause both risks of undertreatment/relapse as well as overtreatment with severe side effects.

In the attempt to achieve individualized 6-mercaptopurine dosing different approaches have been pursued. Nonetheless variation in bioavailability remains a problem.

Earlier, oral tablets of 50 mg (Purinethol) were the only administration form of 6-mercaptopurine and it was primarily designed for adult patients. Challenges with accurate dosing and getting the children to swallow the tablets have been a widespread problem, forcing the caregivers to divide or crush the tablets as well as having to administer different dosages over 2-3 days. Due to these problems, an oral liquid formulation of 6-mercaptopurine (Xaluprine) has been developed. However this oral liquid has only been tested on healthy adult volunteers, and not on the target group, childhood patients. This project will assess the bioavailability and plasma kinetics of oral liquid and tablet formulation of 6-mercaptopurine in children with acute lymphoblastic leukemia.

The investigators hypothesize to observe comparable plasma kinetics, in children with acute lymphoblastic leukemia when treated with 6-mercaptopurine in the form of a tablet and oral liquid formulation, as previously observed in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Childhood acute lymphoblastic leukemia patients, age 0-18 years at diagnosis, treated at the department of pediatrics and adolescent medicine, Rigshospitalet.
* Informed consent

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Time to maximum concentration (Tmax) | Will be measured within a six months after collection of the blood samples
  Time to maximum concentration (Tmax)

SECONDARY OUTCOMES:
Area under curve(AUC) | Will be measured within six months after collection of the blood samples
  Area under curve(AUC)
Maximum concentration (Cmax) | Will be measured within six months after collection of the blood samples
  Maximum concentration (Cmax)
Time to half-life (T½) | Will be measured within six months after collection of the blood samples
  Time to half-life (T½)

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Schmiegelow, Professor, Principal Investigator — Pediatric Clinic II, Rigshospitalet, Copenhagen
Locations (1):
- Juliane Marie Centret, Rigshospitalet, Copenhagen, DK-, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Larsen RH, Hjalgrim LL, Grell K, Kristensen K, Pedersen LG, Brunner ED, Als-Nielsen B, Schmiegelow K, Nersting J. Pharmacokinetics of tablet and liquid formulations of oral 6-mercaptopurine in children with acute lymphoblastic leukemia. Cancer Chemother Pharmacol. 2020 Jul;86(1):25-32. doi: 10.1007/s00280-020-04097-x. Epub 2020 Jun 9. PMID 32519032